CLINICAL TRIAL: NCT06166225
Title: A Remote-based Yoga Intervention for Improving Long-term Weight Loss
Brief Title: Strategies for Improving Remote-based Weight Loss (PATH Trial)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Miriam Hospital (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1947629; R01AT011868 (NIH)
Record Dates: First submitted 2023-12-03; First posted 2023-12-12 (Actual); Last update posted 2025-05-08 (Actual); Status verified 2025-02

CONDITIONS: Obesity
Keywords: yoga; weight loss; exercise; diet
MeSH Terms: conditions — Obesity; Weight Loss; Motor Activity | interventions — Yoga; Health

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Internet-based weight loss program + Iyengar yoga (Experimental): Participants randomized to this group will receive a 12-month automated weight loss program which is delivered via the Internet and will also receive a 9-month Iyengar yoga intervention (delivered during months 4-12). Yoga classes will be delivered live (via Zoom) and participants will be instructed to attend two classes per week for the first 14 weeks and one class per week thereafter. They will also be asked to do self-guided yoga practice on their own and report their yoga practice on the study website.
  Interventions: Behavioral: Internet-based weight loss program; Behavioral: Yoga
- Internet-based weight loss program + health and wellness classes (Active Comparator): Participants randomized to this group will receive a 12-month automated weight loss program which is delivered via the Internet and will also receive a 9-month health and wellness intervention (delivered during months 4-12). Health and wellness classes will be delivered live (via Zoom) and participants will be instructed to attend two classes per week for the first 14 weeks and one class per week thereafter. Classes will consist of lectures, videos, and discussions and will provide education around a variety of lifestyle topics.
  Interventions: Behavioral: Internet-based weight loss program; Behavioral: Health and Wellness

INTERVENTIONS:
Behavioral: Internet-based weight loss program — 12-month, automated and behaviorally-based, Internet-delivered weight loss and weight loss maintenance program
Behavioral: Yoga — 9-month Iyengar yoga program consisting of live (Zoom) yoga classes delivered 1-2 times per week during months 4-12, and self-guided yoga practice recommendations.
  Arms: Internet-based weight loss program + Iyengar yoga
Behavioral: Health and Wellness — 9-month health and wellness program consisting of live (Zoom) yoga classes delivered 1-2 times per week during months 4-12.
  Arms: Internet-based weight loss program + health and wellness classes

SUMMARY:
The purpose of this study is to examine whether the addition of online yoga classes, compared to health and wellness classes, can improve the amount of weight loss produced from an Internet-based weight loss program. All individuals will receive a 12-month, automated Internet-based weight loss program. Following 3 months of of weight loss treatment, individuals will be randomized to also receive yoga classes or health and wellness classes for 9 months. Assessments will occur at baseline, 3, 6, 12, and 18 months and will include measures of weight, eating behaviors, physical activity, and psychosocial factors.

DETAILED DESCRIPTION:
All individuals enrolled in this study will receive a 12-month Internet-based weight loss program, consisting of a 3-month weight loss program, followed by a 9-month weight loss maintenance program. Each week during the first 3 months individuals will be asked to view a 10 to 15-minute multi-media lesson. These lessons focus on behavioral principles for changing diet and physical activity behaviors. Participants are also given weight loss, calorie intake, and physical activity goals. They are taught how to self-monitor this information and are instructed to submit it weekly on the study website. Automated, weekly individualized feedback is provided. Following the 3-month weight loss program participants will receive a 9-month weight loss maintenance program. During this time, they will be asked to view monthly video lessons which focus on strategies for successful weight loss maintenance and be instructed to continue to self-monitor weight, calorie intake, and physical activity minutes on the study website. Automated, monthly feedback is provided.

In addition, participants completing the 3-month weight loss program will be randomly assigned to receive either 9 months of Iyengar yoga classes or 9 months of health and wellness classes. These classes will be held twice per week (live via Zoom) for 14 weeks and then once per week thereafter.

To evaluate the program, participants are asked to complete assessments prior to starting the program (baseline) and at 3, 6, 12 (post-treatment), and 18 months (6 months after completion of the program). For these assessments, participants will be asked to weigh themselves on their study scale, complete a series of online surveys, wear a physical activity monitor for 10 days, and answer daily surveys on their smartphone for 10 days.

ELIGIBILITY:
Inclusion Criteria:

* BMI: 25-40 kg/m2
* Must own smartphone and have daily, home Internet access

Exclusion Criteria:

* Currently pregnant, planning to become pregnant within the next 18 months, or pregnant within the past 6 months
* Current or recent enrollment (<2 years) in a weight loss program
* Current or recent yoga, meditation, or mindfulness practice, either at home or in a studio (defined as ≥12 sessions within the past 2 years)
* Presence of any medical condition for which yoga, exercise, weight loss, or dietary restriction is not recommended
* Recent weight loss (≥10 pounds within the past 6 months)
* Currently taking weight loss medications
* History of bariatric surgery
* Inability to walk 2 blocks without stopping
* Baseline smartphone survey completion rate <80%

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 210 (Estimated)
Dates: Start 2024-01-08 (Actual); Primary Completion 2028-03-30 (Estimated); Study Completion 2028-03-30 (Estimated)

PRIMARY OUTCOMES:
Percent weight change | 12 months
  Weight change will be assessed via smart scales using weight at baseline and 12 months

SECONDARY OUTCOMES:
Dietary lapses | 12 months
  Dietary lapses will be assessed via ecological momentary assessment (EMA). Participants receive EMA surveys 5x/day, for 10 days, at baseline and 12 months, and surveys ask about any dietary lapses since completing the last survey.
Affect | 12 months
  Affect will be assessed via ecological momentary assessment (EMA). Participants receive EMA surveys 5x/day, for 10 days, at baseline and 12 months, and surveys ask about current affect.
Dietary temptations | 12 months
  Dietary temptations will be assessed via ecological momentary assessment (EMA). Participants receive EMA surveys 5x/day, for 10 days, at baseline and 12 months, and surveys ask about dietary temptations experienced since the last prompt.
Percentage of time that tempting foods were eaten | 12 months
  Dietary temptations will be assessed via ecological momentary assessment (EMA). Participants receive EMA surveys 5x/day, for 10 days, at baseline and 12 months, and surveys ask about dietary temptations experienced since the last prompt. If a temptation is reported, participants are asked to state whether they ate the tempting food. The percentage of time that tempting foods were eaten (vs. not eaten) will be calculated.
Dispositional mindfulness | 12 months
  Mindfulness will be assessed via the Five Facet Mindfulness Questionnaire - Short Form at baseline and 12 months
Distress tolerance | 12 months
  Distress tolerance will be assessed via the Distress Tolerance Scale at baseline and 12 months
Self-compassion | 12 months
  Self-compassion will be assessed via the Self-Compassion Scale - Short Form at baseline and 12 months
Behavioral inhibition | 12 months
  Behavioral inhibition will be assessed via the Behavioral Inhibition System and Behavioral Activation System (BIS/BAS) Questionnaire at baseline and 12 months and the BIS subscale will be assessed.
Self-efficacy | 12 months
  Self-efficacy will be assessed using the Weight Efficacy Lifestyle Questionnaire at baseline and 12 months.

OTHER OUTCOMES:
Percent weight change | 18 months
  Weight change will be assessed via smart scales using weight at baseline and 18 months to examine the long-term effects of the interventions.

CONTACTS AND LOCATIONS:
Locations (1):
- The Miriam Hospital's Weight Control and Diabetes Research Center, Providence, Rhode Island, United States

IPD SHARING:
Plan to Share IPD: Yes
Data will available to other researchers as raw individual-level data; however, this will not be available until the primary outcome papers from the study are accepted for publication. Requestors will be required to sign a data sharing agreement stating that: (1) They will use the data for research purposes only unless otherwise agreed, and will not identify any individual or personal information, (2) Data will be secured using appropriate technology/firewalls, (3) Data will be destroyed after data analysis, and (4) They will cite data appropriately in publications or other written materials. A record of transfer of data and a copy of the dataset that was distributed will be kept by The Miriam Hospital
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Study data will be made available as soon as possible, but no later than within one year of the completion of the funded project period or upon acceptance of the data for publication.